CLINICAL TRIAL: NCT00732290
Title: Investigation of Drug-drug Interaction Between Clopidogrel and Fluoxetine
Acronym: PLATINE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 0801068; 2008-004395-46
Record Dates: First submitted 2008-08-08; First posted 2008-08-11 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-03

CONDITIONS: Healthy
Keywords: Healthy volunteer; Pharmacokinetic; pharmacodynamic; Polymorphism, Genetic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Clopidogrel then fluoxetine+clopidogrel
  Interventions: Drug: Clopidogrel then fluoxetine+clopidogrel
- 2 (Active Comparator): Fluoxetine+clopidogrel then clopidogrel
  Interventions: Drug: Fluoxetine+clopidogrel then clopidogrel

INTERVENTIONS:
Drug: Clopidogrel then fluoxetine+clopidogrel — D1 : clopidogrel (Plavix) 600mg (8 tablets) one time D45 to D48 : Fluoxetine (Fluoxetine EG 20mg) 20mg (1 tablet) per day D49 : 20mg Fluoxetine + 600mg Clopidogrel
  Arms: 1
Drug: Fluoxetine+clopidogrel then clopidogrel — D1 to D4 : Fluoxetine (Fluoxetine EG 20mg) 20mg (1 tablet) per day D5: 20mg Fluoxetine + Clopidogrel (Plavix) 600mg (8 tablets) one time D49 : Clopidogrel 600mg one time
  Arms: 2

SUMMARY:
Clopidogrel is a platelet aggregation inhibitor witch prevents thrombotic events in patients with atherosclerotic vascular disease. To date, 4 to 30 % of patients are considered as poor, low or non-responder to this therapeutic. However, drug-drug interactions may lead to decrease the clopidogrel responsiveness. Many arguments are in support to a drug-drug interaction between clopidogrel and fluoxetine (selective serotonin reuptake inhibitor). On the pharmacokinetic level, fluoxetine inhibits the cytochroms involved in the production of clopidogrel active metabolite. On the pharmacodynamic level fluoxetine could increase the risk of hemorrhage by inhibiting the serotonin platelet reuptake and thus enhance the antiplatelet effect of clopidogrel.

The purpose of this study is to investigate the influence of fluoxetine on pharmacokinetic and pharmacodynamic of clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

* Signed an informed consent
* Body mass: 60 to 85 Kg
* Platelet count: 180 to 350 G/L
* % platelet aggregation > 70%
* Subjects are to be in good health as determined by a medical history, physical examination including vital signs, and clinical laboratory test results including liver function, renal and full blood count

Exclusion Criteria:

* Subject with an history of seizure disorder
* Subject with a known allergy fluoxetine or clopidogrel
* Cigarette smoking
* Subject with a history of hemorrhagic disease
* Peptic ulcer
* Psychiatric disorders
* Participation in another clinical or device trial within the three previous months
* Subject who is currently taking medications
* Subject who is currently taking medications for depression
* Subject with an history of depression (MADRS score < 15)
* Hepatic insufficiency

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Platelet aggregation inhibition measured by optical aggregometry in presence of adenosine diphosphate (ADP) 20 μmol/L and 5 μmol/L. | Before first fluoxetin taking, during clopidogrel taking

SECONDARY OUTCOMES:
Level of phosphorylated VASP (vasodilator- stimulated phosphoprotein), a good index of P2Y12 activity (platelet receptor of clopidogrel) and P-selectin by flow cytometry. | Before first Fluoxetine taking and during Clopidogrel taking
Determination of clopidogrel and its metabolites in plasma by LC/MS-MS method | During clopidogrel taking

CONTACTS AND LOCATIONS:
Overall Officials: Pierre GARNIER, MD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- Service de Medecin et Therapeutique, Unite de Recherche Clinique Groupe de Recherche sur la Thrombose (EA3065), Saint-Etienne, France